CLINICAL TRIAL: NCT02024945
Title: Evaluation of Health-Related Quality of Life in Patients With Overactive Bladder Syndrome (OAB) Treated With Propiverine, and Its Efficacy and Tolerance in Daily Practice in Belgian General Practitioners and Urologists
Brief Title: Efficacy, Tolerability and Impact on Quality of Life of Propiverine in Patients With Overactive Bladder Syndrome
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: MN-9999-401-BE; U1111-1146-5884 (Other: World Health Organization)
Record Dates: First submitted 2013-12-28; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Overactive Bladder Syndrome
Keywords: Drug therapy
MeSH Terms: interventions — propiverine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Propiverine: Participants with symptoms of OAB, prescribed propiverine in accordance with the summary of product characteristics (SPC).
  Interventions: Drug: Propiverine

INTERVENTIONS:
Drug: Propiverine — Propiverine 15 mg tablets or 30 mg regulated release capsules
  Other Names: Mictonorm®; Mictonorm Uno®

SUMMARY:
The purposes of this study were to assess Quality of Life (QoL) and urination urge, incontinence, and micturition frequency including nocturia after 4 and 12 weeks treatment with propiverine.

DETAILED DESCRIPTION:
The drug being tested in this study is called propiverine. Propiverine is being tested to evaluate Quality of Life (QoL) and improvement of OAB symptoms in people who take propiverine. The study will enroll approximately 1000 patients who the treating physician decided to treat with propiverine 15mg tablets or 30 mg regulated release capsules as part of their normal clinical practice. All participants will be asked to keep a voiding diary for 2 consecutive days and to complete a QoL questionnaire after 1st visit and before each subsequent visit. This multi-centre trial will be conducted in Belgium. The overall time to participate in this study is up to 12 weeks. Participants will make 3 visits to their healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent. 2. At least 18 years of age. 3. Patients with complaints of Overactive Bladder Syndrome (OAB) without urge incontinence, OAB with urge incontinence, or with mixed urinary incontinence. 4. Patients who consult their GP or an urologist for the first time with these complaints or who stopped their OAB treatment since at least one month. 5. Receiving a propiverine prescription according to the Summary of Product Characteristics (SPC).

Exclusion Criteria:

* None, as per the SPC contra-indications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OAB symptoms, who the treating physician decided to treat with propiverine, were to be included by General Practitioners (GP) and urologists in private practice in Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Quality of Life (QoL) as assessed by the King's Health Questionnaire (KHQ) at Weeks 4 and 12 | Baseline, Weeks 4 and 12
  The King's Health Questionnaire is a condition-specific health-related QoL instrument for the assessment of patients with lower urinary tract conditions including overactive bladder. It is a self-administered questionnaire containing 21 questions scored in 9 domains (general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep or energy, and severity of urinary symptoms). All domains were assessed in a range: 0-100, where 0=best and 100=worst outcome. Lower scores indicates better QoL.
Change from Baseline in Urination Urge at Weeks 4 and 12 | Baseline, Weeks 4 and 12
  Each participant kept a voiding diary and recorded urinary urgency. The diary was kept for 2 consecutive days within 7 days of the Baseline visit, and 2 consecutive days just before the Week 4 and 12 visits. The average urination urge was then calculated.
Change from Baseline in Incontinence episodes at Weeks 4 and 12 | Baseline, Weeks 4 and 12
  Each patient kept a voiding diary and episodes of incontinence. The diary was kept for 2 consecutive days within 7 days of the Baseline visit, and 2 consecutive days just before the Week 4 and 12 visits. The average number of incontinence episodes per 24 hours was calculated.
Change from Baseline in Micturition Frequency including nocturia at Weeks 4 and 12 | Baseline, Weeks 4 and 12
  Each patient kept a voiding diary and recorded the number of micturitions. The diary was kept for 2 consecutive days within 7 days of the Baseline visit, and 2 consecutive days just before the Week 4 and 12 visits. The average number of micturitions and nocturia episodes per 24 hours was calculated.

SECONDARY OUTCOMES:
Change from Baseline in Urine Volume per Void at Weeks 4 and 12 | Baseline, Weeks 4 and 12
  Mean volume per void (or amount of urine per urination) over 24 hours is based on a 2-day diary maintained by the participant.
Patient and Investigator Assessment of Efficacy of Propiverine at Weeks 4 and 12 | Weeks 4 and 12
  Evaluation of efficacy was assessed by participants and investigators on a 4 point scale. Participants and investigators reported efficacy as very good, good, sufficient, or insufficient.
Patient and Investigator Assessment of Tolerability of Propiverine at Weeks 4 and 12 | 12 Weeks
  Evaluation of tolerability was assessed by participants and investigators on a 4 point scale. Participants and investigators reported tolerability as very good, good, sufficient, or insufficient.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda